CLINICAL TRIAL: NCT03893058
Title: Evaluation of the NeuroMuscular Junction Using the Single Fiber Electromyography and Reliability of Train-Of-Four in Critically Ill Patients.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Matteo Filippini, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: NP2963
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Critical Illness Polyneuropathy; Critical Illness Myopathy; Weakness Due to Disease; Neuromuscular Blockade
Keywords: Train-Of-Four; Single Fiber Electromyography; NeuroMuscular Junction; Critical Illness
MeSH Terms: conditions — Polyneuropathies; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients suffering from critical illnesses who are admitted to the Intensive Care Unit (ICU) are often affected by multiple organ failure. Among those dysfunctions, it is very important to mention the neuromuscular system failure, known as Intensive Care Unit-Acquired Weakness (ICU-AW). In non-cooperative patients, the simplified electromyography (called Peroneal Nerve Test, PENT) allows diagnosing the Critical Illness Polyneuropathy (CIP) and/or the Critical Illness Myopathy (CIM), which are two causes of ICU-AW. The ICU-AW can involve both nerves and muscles, but so far there has been no evidence about the involvement of the third element of the neuromuscular system: the neuromuscular junction (NMJ). The gold standard technique to study the function of the NMJ is the Desmedt test, a particular type of Electroneurography (ENG); the Single Fiber Electromyography (SF-EMG ) might be a valid and more sensitive technique for this analysis. The spreading use of Neuromuscular Blocking Agents (NMBAs) has led to the introduction of the Train-Of-Four acceleromyography (TOF) monitoring in ICU; however, there is a lack of information on its reliability in critically ill patients.

Some conditions related to critical illness, like the ICU-AW, could make TOF monitoring unreliable.

The aims of the study are:

1. To estimate the prevalence of NMJ disorders acquired during critical illnesses using SF-EMG.
2. To assess the reliability of TOF in critically ill patients. The study will evaluate patients with critical illnesses hospitalised in the General Intensive Care Unit (UOC Anestesia e Rianimazione 2, Spedali Civili di Brescia). To diagnose CIP and/or CIM, PENT will be performed after 72 hours from the admission in the ICU and every 72 hours. To evaluate NMJ disorders, SF-EMG will be performed in patients with an abnormal PENT. To evaluate the reliability of TOF, the test will be performed before, during and after NMBAs treatment and in all studied patients, independently from NMBAs administration; the presence of neuromuscular blockade will be evaluated clinically and/or using instrumental tests like Desmedt test. Statistical analysis will be performed to represent the prevalence of NMJ disorders in the general intensivistic population and the reliability of TOF in terms of specificity and sensitivity for the diagnosis of the neuromuscular blockade.

DETAILED DESCRIPTION:
COMPLETE TITLE OF THE STUDY: EVALUATION OF THE NEUROMUSCULAR JUNCTION USING THE SINGLE FIBER ELECTROMYOGRAPHY AND RELIABILITY OF TRAIN-OF-FOUR IN CRITICALLY ILL PATIENTS. Author and responsible for the study: Dr. Matteo Filippini Sponsor: ASST Spedali Civili di Brescia - Italy

1. RATIONALE OF THE STUDY Patients suffering from critical illnesses who are admitted to the Intensive Care Unit (ICU) are often affected by multiple organ failure. Among those dysfunctions, it is very important to mention the neuromuscular system failure, known as Intensive Care Unit-Acquired Weakness (ICU-AW). In non-cooperative patients, the simplified electromyography (called Peroneal Nerve Test, PENT) allows diagnosing the Critical Illness Polyneuropathy (CIP) and/or the Critical Illness Myopathy (CIM), which are two causes of ICU-AW. The ICU-AW can involve both nerves and muscles, but so far there has been no evidence about the involvement of the third element of the neuromuscular system: the neuromuscular junction (NMJ). The gold standard technique to study the function of the NMJ is the Desmedt test, a particular type of Electroneurography (ENG); the Single Fiber Electromyography (SF-EMG ) might be a valid and more sensitive technique for this analysis. The spreading use of Neuromuscular Blocking Agents (NMBAs) has led to the introduction of the Train-Of-Four acceleromyography (TOF) monitoring in ICU; however, there is a lack of information on its reliability in critically ill patients. Some conditions related to critical illness, like the ICU-AW, could make TOF monitoring unreliable.
2. STUDY AIMS A. To estimate the prevalence of NMJ disorders acquired during critical illnesses using SF-EMG. B. To assess the reliability of TOF in critically ill patients.
3. POPULATION Target population: patients with critical illnesses hospitalised in the General Intensive Care Unit (UOC Anestesia e Rianimazione 2, Spedali Civili di Brescia). Inclusion criteria: adult patients (18-year-old and older ones) hospitalised in ICU. In order to realise the first aim of the study, patients with a pathologic PENT will be evaluated. In order to realise the second aim of the study, patients who receive NMBAs will be evaluated; patients who do not receive NMBAs will also be evaluated, as a control group.

   Exclusion criteria:
   * patients with a terminal disease;
   * patients with an ICU-length-of-staying perspective less than 72 hours;
   * patients with a chronic disease associated with known neuropathy or myopathy;
   * patients treated with drugs that may cause neurotoxicity and myotoxicity;
   * patients with primary or secondary acute Peripheral Nervous System (PNS) lesions or muscle lesions;
   * patients with prosthesis, wounds or other conditions that prevent electrophysiological testing.
4. STUDY DESIGN Observational, prospective, cohort study; retrospective analysis of prospectively collected data.
5. OPERATIVE PROCEDURES

   * to diagnose CIP and/or CIM, PENT will be performed after 72 hours from the admission in the ICU and every 72 hours.
   * to evaluate NMJ disorders, SF-EMG will be performed in patients with an abnormal PENT.
   * to evaluate the reliability of TOF, the test will be performed before, during and after NMBAs treatment and in all studied patients, independently from NMBAs administration; the presence of the neuromuscular blockade will be evaluated clinically and/or using instrumental tests like Desmedt test.

   PROCEDURES:

   SIMPLIFIED ELECTROMYOGRAPHY (EMG) The simplified EMG is called Peroneal Nerve Test (PENT), and it consists in measuring the compound muscle action potential (CMAP) of a single peroneal nerve (if the first peroneal nerve tested is pathologic) or of both peroneal nerves (if the first nerve is healthy). ICU-AW is diagnosed in case of reduction of CMAP under the usual cutoff (calculated as two standard deviations from the average laboratory value). SF-EMG - SINGLE FIBER ELECTROMYOGRAPHY The Single Fiber Electromyography (SF-EMG) is a test which studies action potentials of single muscular fibre. It allows the study of muscular fibres microphysiology, and it investigates early alterations (sometimes preclinical) of NMJ, typical of Myasthenia Gravis. The needle electrode for the single fibre analysis is composed of a small registration surface, and this is the cathode, while a second electrode is the anode. The muscle action potential registration follows the tested muscles activation and this activation can be voluntary (voluntary SF-EMG) or through stimulation (stimulated SF-EMG), with a stimulation frequency of 2-10 Hz, an intensity of 10-20 mA and a duration between 10-50 ms. The variation in the time interval between two action potentials of the same motor unit is called "jitter". SF-EMG measures the variation of this inter potential interval (jitter), which can be increased in patients with NMJ diseases. TOF - TRAIN-OF-FOUR ACCELEROMYOGRAPHY The TOF acceleromyography consists in the consecutive application of four electrical stimuli (generally 200 ms, 50 mA) through the course of the ulnar nerve and in the recording of the induced thumb acceleration; the result of this test is expressed as the ratio of the fourth to the first magnitude of the response. If the ratio is greater than 90%, the response will be considered normal, and the clinical meaning of this finding is that the patient is not (or no more) under the effect of NMBAs. Conversely, if the ratio is less than 90%, the clinical meaning is that the patient is under the effect of non-depolarising NMBAs. TOOLS Paper and electronic detection boards. OTHER EVALUATIONS Collection of clinical data useful for describing the status of the investigated population. DATA MANAGEMENT Electrophysiological measurements data conducted to the patient's bed will be integrated with clinical-physical and laboratory data ordered in a worksheet (progressive number, diagnosis, initials, age, sex, weight, height, BMI, days of hospitalization, length of staying in the ICU, previous surgical procedures, inflammation indexes, liver and kidney function indexes, coagulation function indexes, mechanical ventilation mode, simplified acute physiology score II [SAPS II] and sequential order failure assessment [SOFA] score). Data collection: data will be collected daily by the principal investigator, as well as by students and resident physicians involved in the project and previously provided with appropriate authorisation to attend the centre for training purposes. Rules on personal data management: see the next point for the respect of privacy. Operational methods of data management: recording of data on paper and/or electronic card without uploading to file, management of electronic archives or linkage procedures with other databases.
6. STATISTICAL ANALYSIS AND METHODS

   A descriptive statistical analysis will be performed to represent:

   A. The characteristics of the population: number of subjects, sex, age, body mass index (BMI), Glasgow Come Score (GCS), SOFA score and SAPS II, days of hospitalization in ICU, reason for admission to ICU, use of amines, presence and severity of the infectious state. In particular:
   * Qualitative variables (e.g. sex, disease) will be expressed as mode and frequency distribution.
   * Ordinal quantitative variables (e.g. GCS) will be expressed as median and interquartile range.
   * Continuous quantitative variables (e.g. age, BMI) will be expressed as mean and standard deviation.

   B. The results of the applied diagnostic tests:
   * the result of the PENT will be expressed as the magnitude of the potential (mV);
   * the result of the SF-EMG will be expressed as the variation in the time interval between the two action potentials of the same motor unit (jitter) (msec)
   * the result of the TOF will be expressed as the ratio of the fourth response magnitude to the first one. An inferential statistical analysis will be performed to represent the prevalence of NMJ disorders in the general intensivistic population and the reliability of TOF in terms of specificity and sensitivity for the diagnosis of the neuromuscular blockade. SAMPLE SIZE The investigator's hypothesis is that NMJ disorders in the study population are non-existent or in any case epidemiologically irrelevant: therefore a sample of 73 patients with a negative test will allow affirming that the prevalence of that disorder is less than 10%. If one or more SF-EMG tests are positive, the prevalence of NMJ disorders will be calculated from those results with a 95% confidence interval. After the enrolment of 35 patients studied with SF-EMG, an ad-interim analysis will be performed, and the prevalence of NMJ disorders will be estimated by an exact binomial test, and the 95% confidence interval will be calculated. In order to realise the second aim of the study (to assess the reliability of TOF in critically ill patients) a sample of 85 patients will allow estimating sensitivity and specificity with a precision of 10% under the realistic hypothesis that they are 100% and 90% respectively.
7. ETHICAL ASPECTS The study, being observational, will not entail, in itself, any risk for any patient. The data of the patients included in the study will be physical-technical (PENT and SF-EMG tests) and clinical-laboratoristic. They will be obtained from standard clinical practice. The investigator will proceed to exhaustive information about the nature of the study and the operations of analysis towards patients; the same patients, made aware of the nature of the collected data, will be required to express the informed consent, according to the regulations in force. In the case of patients unable to give valid consent, data collection and processing will only take place after the patients themselves have regained their lost capacity and have given consent or after this has been done by legal representatives. The study does not alter the risk/benefit ratio of the procedures used for data acquisition; concerning the specific acts of the study, this ratio is zero. This study will be conducted in accordance with this protocol, with the principles of good clinical practice in accordance with the International Conference on Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH GCP) guidelines and ethical principles set out in the Helsinki Declaration.
8. INFORMATION TO THE PATIENT AND CONSENT The patients will express their informed consent to the conduct of the study and the management of sensitive data by signing their own form on the specially prepared forms. In the case of patients lacking the ability to act and for which there is a legal representative, the informed consent will be given by the latter. The informative note before the acquisition of consent will be provided by the principal investigator.
9. APPROVAL BY THE RESPONSIBLE ETHICS COMMITTEE The documents of the study were reviewed and approved by the responsible Ethics Committee (Comitato Etico di Brescia, NP2963).
10. CONFIDENTIALITY OF DATA AND PRIVACY The confidentiality of the collected data (including laboratory data) will be maintained through the rigorous conservation of data collection cards by the investigators and the patients involved will be identified with codes that guarantee anonymity, even in order to comply with the privacy of the subjects, according to the law in force.
11. DATA PROPERTY The ownership of the data related to the study, its execution and its results belong to the sponsor.
12. PUBLICATION OF RESULTS The investigator reserves the right to publish the results of the study through works published in specialised journals whose editorial policies respect the laws in force, with particular reference to the anonymity of the data.
13. CONSERVATION OF STUDY DOCUMENTS All information related to the study participants, including data collection forms, documentation "source" (in addition to the medical records already stored by the hospital), all clinical and laboratory data used for the study, as well as all the documentation concerning the submission and approval by the Ethics Committee, the informed consent and all the regulatory documentation, etc. will be kept by the investigators in a safe and accessible place for possible inspections.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (18-year-old and older ones) hospitalised in ICU. In order to realise the first aim of the study (to estimate the prevalence of NMJ disorders acquired during critical illnesses using SF-EMG), patients with a pathologic PENT will be evaluated. In order to realise the second aim of the study (to assess the reliability of TOF in critically ill patients. The study will evaluate patients with critical illnesses hospitalised in the General Intensive Care Unit), patients who receive NMBAs will be evaluated; patients who do not receive NMBAs will also be evaluated, as a control group.

Exclusion Criteria:

* patients with a terminal disease;
* patients with an ICU-length-of-staying perspective less than 72 hours;
* patients with a chronic disease associated with known neuropathy or myopathy;
* patients treated with drugs that may cause neurotoxicity and myotoxicity;
* patients with primary or secondary acute Peripheral Nervous System (PNS) lesions or muscle lesions;
* patients with prosthesis, wounds or other conditions that prevent electrophysiological testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with critical illnesses hospitalised in the General Intensive Care Unit (UOC Anestesia e Rianimazione 2, Spedali Civili di Brescia)
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NeuroMuscularJunction disorders acquired during critical illnesses. | 3 years
  The prevalence will be assessed as the proportion of patients found to be affected by NMJ disorders (assessed by SFEMG) among the population of critically ill patients.
Reliability (specificity and sensitivity) of Train-Of-Four in critically ill patients. | 3 years
  The sensitivity of TOF for the diagnosis of the neuromuscular blockade will be expressed as the proportion of patients with the neuromuscular blockade and with abnormal TOF ratio (<90%) among patients with the neuromuscular blockade and with normal or abnormal TOF ratio.
  The specificity of TOF for the diagnosis of the neuromuscular blockade will be expressed as the proportion of patients without the neuromuscular blockade and with normal TOF ratio (>90%) among patients without neuromuscular blockade and with normal or abnormal TOF ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farhan H, Moreno-Duarte I, Latronico N, Zafonte R, Eikermann M. Acquired Muscle Weakness in the Surgical Intensive Care Unit: Nosology, Epidemiology, Diagnosis, and Prevention. Anesthesiology. 2016 Jan;124(1):207-34. doi: 10.1097/ALN.0000000000000874. PMID 26445385
- [Background] Argov Z, Latronico N. Neuromuscular complications in intensive care patients. Handb Clin Neurol. 2014;121:1673-85. doi: 10.1016/B978-0-7020-4088-7.00108-5. PMID 24365440
- [Background] Eikermann M, Latronico N. What is new in prevention of muscle weakness in critically ill patients? Intensive Care Med. 2013 Dec;39(12):2200-3. doi: 10.1007/s00134-013-3132-4. Epub 2013 Oct 24. No abstract available. PMID 24154675
- [Background] Latronico N, Filosto M, Fagoni N, Gheza L, Guarneri B, Todeschini A, Lombardi R, Padovani A, Lauria G. Small nerve fiber pathology in critical illness. PLoS One. 2013 Sep 30;8(9):e75696. doi: 10.1371/journal.pone.0075696. eCollection 2013. PMID 24098716
- [Background] Latronico N, Tomelleri G, Filosto M. Critical illness myopathy. Curr Opin Rheumatol. 2012 Nov;24(6):616-22. doi: 10.1097/BOR.0b013e3283588d2f. PMID 22918529
- [Background] Latronico N, Bolton CF. Critical illness polyneuropathy and myopathy: a major cause of muscle weakness and paralysis. Lancet Neurol. 2011 Oct;10(10):931-41. doi: 10.1016/S1474-4422(11)70178-8. PMID 21939902
- [Background] Latronico N, Rasulo FA. Presentation and management of ICU myopathy and neuropathy. Curr Opin Crit Care. 2010 Apr;16(2):123-7. doi: 10.1097/MCC.0b013e328336a229. PMID 20075723
- [Background] Katirji B, Kaminski HJ. Electrodiagnostic approach to the patient with suspected neuromuscular junction disorder. Neurol Clin. 2002 May;20(2):557-86, viii. doi: 10.1016/s0733-8619(01)00012-3. PMID 12152447
- [Background] Sonoo M, Uesugi H, Mochizuki A, Hatanaka Y, Shimizu T. Single fiber EMG and repetitive nerve stimulation of the same extensor digitorum communis muscle in myasthenia gravis. Clin Neurophysiol. 2001 Feb;112(2):300-3. doi: 10.1016/s1388-2457(00)00544-7. PMID 11165533
- [Background] Padua L, Caliandro P, Di Iasi G, Pazzaglia C, Ciaraffa F, Evoli A. Reliability of SFEMG in diagnosing myasthenia gravis: sensitivity and specificity calculated on 100 prospective cases. Clin Neurophysiol. 2014 Jun;125(6):1270-3. doi: 10.1016/j.clinph.2013.11.005. Epub 2013 Nov 15. PMID 24296278
- [Background] Tschida SJ, Hoey LL, Vance-Bryan K. Inconsistency with train-of-four monitoring in a critically ill paralyzed patient. Pharmacotherapy. 1995 Jul-Aug;15(4):540-5. PMID 7479211
- [Background] Rudis MI, Guslits BG, Zarowitz BJ. Technical and interpretive problems of peripheral nerve stimulation in monitoring neuromuscular blockade in the intensive care unit. Ann Pharmacother. 1996 Feb;30(2):165-72. doi: 10.1177/106002809603000211. PMID 8835051
- [Background] Lagneau F, Benayoun L, Plaud B, Bonnet F, Favier J, Marty J. The interpretation of train-of-four monitoring in intensive care: what about the muscle site and the current intensity? Intensive Care Med. 2001 Jun;27(6):1058-63. doi: 10.1007/s001340100964. PMID 11497139
- [Background] Greenberg SB, Vender J. The use of neuromuscular blocking agents in the ICU: where are we now? Crit Care Med. 2013 May;41(5):1332-44. doi: 10.1097/CCM.0b013e31828ce07c. PMID 23591211
- [Background] Puthucheary Z, Rawal J, Ratnayake G, Harridge S, Montgomery H, Hart N. Neuromuscular blockade and skeletal muscle weakness in critically ill patients: time to rethink the evidence? Am J Respir Crit Care Med. 2012 May 1;185(9):911-7. doi: 10.1164/rccm.201107-1320OE. PMID 22550208
- [Background] Strange C, Vaughan L, Franklin C, Johnson J. Comparison of train-of-four and best clinical assessment during continuous paralysis. Am J Respir Crit Care Med. 1997 Nov;156(5):1556-61. doi: 10.1164/ajrccm.156.5.9701079. PMID 9372675
- [Background] Dieye E, Minville V, Asehnoune K, Conil C, Georges B, Cougot P, Fourcade O, Conil JM. Pharmacodynamics of cisatracurium in the intensive care unit: an observational study. Ann Intensive Care. 2014 Feb 11;4(1):3. doi: 10.1186/2110-5820-4-3. PMID 24521394
- [Background] Latronico N, Nattino G, Guarneri B, Fagoni N, Amantini A, Bertolini G; GiVITI Study Investigators. Validation of the peroneal nerve test to diagnose critical illness polyneuropathy and myopathy in the intensive care unit: the multicentre Italian CRIMYNE-2 diagnostic accuracy study. F1000Res. 2014 Jun 11;3:127. doi: 10.12688/f1000research.3933.3. eCollection 2014. PMID 25309729
- [Background] Latronico N, Gosselink R. A guided approach to diagnose severe muscle weakness in the intensive care unit. Rev Bras Ter Intensiva. 2015 Jul-Sep;27(3):199-201. doi: 10.5935/0103-507X.20150036. Epub 2015 Sep 15. No abstract available. PMID 26376161
- [Background] Fan E, Cheek F, Chlan L, Gosselink R, Hart N, Herridge MS, Hopkins RO, Hough CL, Kress JP, Latronico N, Moss M, Needham DM, Rich MM, Stevens RD, Wilson KC, Winkelman C, Zochodne DW, Ali NA; ATS Committee on ICU-acquired Weakness in Adults; American Thoracic Society. An official American Thoracic Society Clinical Practice guideline: the diagnosis of intensive care unit-acquired weakness in adults. Am J Respir Crit Care Med. 2014 Dec 15;190(12):1437-46. doi: 10.1164/rccm.201411-2011ST. PMID 25496103
- [Background] Latronico N, Bertolini G, Guarneri B, Botteri M, Peli E, Andreoletti S, Bera P, Luciani D, Nardella A, Vittorielli E, Simini B, Candiani A. Simplified electrophysiological evaluation of peripheral nerves in critically ill patients: the Italian multi-centre CRIMYNE study. Crit Care. 2007;11(1):R11. doi: 10.1186/cc5671. PMID 17254336
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Cominotti S, Chiaranda M, Mascetti P, Lucchini E, Severgnini P. [Comparison of SAPS II, MPM II24 and SAPS in intensive care]. Minerva Anestesiol. 1999 Oct;65(10):717-23. Italian. PMID 10598429
- [Background] Unterbuchner C, Blobner M, Puhringer F, Janda M, Bischoff S, Bein B, Schmidt A, Ulm K, Pithamitsis V, Fink H. Development of an algorithm using clinical tests to avoid post-operative residual neuromuscular block. BMC Anesthesiol. 2017 Aug 4;17(1):101. doi: 10.1186/s12871-017-0393-4. PMID 28778151
- [Background] Naguib M, Brull SJ, Johnson KB. Conceptual and technical insights into the basis of neuromuscular monitoring. Anaesthesia. 2017 Jan;72 Suppl 1:16-37. doi: 10.1111/anae.13738. PMID 28044330
- [Background] Buderer NM. Statistical methodology: I. Incorporating the prevalence of disease into the sample size calculation for sensitivity and specificity. Acad Emerg Med. 1996 Sep;3(9):895-900. doi: 10.1111/j.1553-2712.1996.tb03538.x. PMID 8870764